CLINICAL TRIAL: NCT06252064
Title: Rehabilitative Therapy and Pridinol in Patients With Lumbar Spondylarthrosis and Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Prof.ssa Giulia Letizia Mauro, Professor, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MFR022024
Record Dates: First submitted 2024-01-22; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Spondyloarthropathy
Keywords: Spondylarthropathies; Pridinol Mesilate; Low Back Pain; Rehabilitation; Therapy
MeSH Terms: conditions — Spondylarthropathies; Low Back Pain | interventions — Rehabilitation; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Combo Group (Active Comparator): Rehabilitation treatment combined with drug therapy
  Interventions: Other: Rehabilitation + Drug therapy
- Reha Group (Active Comparator): Rehabilitation treatment
  Interventions: Other: Rehabilitation
- Drug Group (Active Comparator): Drug therapy with Pridinol Mesylate
  Interventions: Other: Drug therapy

INTERVENTIONS:
Other: Rehabilitation + Drug therapy — Patients in the Combo group underwent rehabilitation treatment combined with drug therapy: the rehabilitation protocol included daily sessions, 5 days a week, lasting 60 minutes, for a total of 4 consecutive weeks. Patients included in this group also took drug therapy, particularly Pridinol Mesylate orally, on an empty stomach, 2 mg x 3 times a day for 20 days.
  Arms: Combo Group
Other: Rehabilitation — Patients in the Reha group underwent rehabilitation treatment: the rehabilitation protocol included daily sessions, 5 days a week, lasting 60 minutes, for a total of 4 consecutive weeks. The treatment included an initial step, lasting 40 minutes, of Postural Reeducation ending with Stretching exercises of the posterior kinetic chain muscles lasting 20 minutes.
  Arms: Reha Group
Other: Drug therapy — The Drug Group had taken Pridinol Mesylate orally, on an empty stomach, 2 mg x 3 times a day for 20 days. The tablet was taken without chewing and with a glass of water (200 ml). The drug was taken in environments with temperature below 25° C.
  Arms: Drug Group

SUMMARY:
Spondyloarthrosis is a degenerative disease involving the intervertebral disc, vertebral bodies, and adjacent soft tissues. Treatment aims to slow disease progression and manage symptoms through an interdisciplinary approach.It can be conservative, pharmacological and interventional, rarely chirurgic. This study aimed to evaluate the effectiveness of a rehabilitation program combined with Pridinol Mesylate in the treatment of Spondyloarthrosis in elderly patients in terms of pain resolution, improving disability, and quality of life versus single treatment.

A randomized controlled trial was conducted in patients with spondyloarthritis. The patients recruited were divided into three groups: the Combined Group (CG), who received a rehabilitation program combined with Pridinol Mesylate; the Rehabilitation Group (RG), who received only the same rehabilitation program; and the Drug Group (DG), who received only the administration of the drug.

ELIGIBILITY:
Inclusion Criteria:

* age 65-75 years,
* low back pain for at least 3 months,
* NRS ≥ 4,
* radiographic diagnosis of spondyloarthrosis,
* written informed consent.

Exclusion Criteria:

* inflammatory diseases of the spine,
* obesity (BMI 20-30),
* positive radicular tests,
* allergy or contraindications related to taking Pridinol Mesylate.

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 86 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Extent of pain: Numeric Rating Scale (NRS 0-10) | at recruitment (T0), after 20 days of treatment (T1), after 90 days from recruitment (T2)
  The NRS is a subjective scale that rates the extent of pain with a score between 0 and 10; a score of 10 corresponds to maximum pain.

SECONDARY OUTCOMES:
Quality of life: Short Form Health Survey 36 (0-100) | at recruitment (T0), after 20 days of treatment (T1), after 90 days from recruitment (T2)
  SF-36 is a scale that assesses the quality of life in relation to the disease from which patients suffer. A score of 100 corresponds to an optimal value.
Disability: Quebec Back Pain Disability Scale (QBPDS scale 0-100) | at recruitment (T0), after 20 days of treatment (T1), after 90 days from recruitment (T2)
  is a condition-specific questionnaire developed to measure the level of functional disability for patients with low back pain. These outcomes score within the range of 0 and 100, determents the level of functional disability, with higher numbers representing greater levels of disability.

CONTACTS AND LOCATIONS:
Overall Officials: Giulia Letizia Mauro, Principal Investigator — A.O.U.P. Paolo Giaccone Palermo
Locations (1):
- Functional Recovery and Rehabilitation Unit of the A.O.U.P. Paolo Giaccone, Palermo, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Qaseem A, Wilt TJ, McLean RM, Forciea MA; Clinical Guidelines Committee of the American College of Physicians; Denberg TD, Barry MJ, Boyd C, Chow RD, Fitterman N, Harris RP, Humphrey LL, Vijan S. Noninvasive Treatments for Acute, Subacute, and Chronic Low Back Pain: A Clinical Practice Guideline From the American College of Physicians. Ann Intern Med. 2017 Apr 4;166(7):514-530. doi: 10.7326/M16-2367. Epub 2017 Feb 14. PMID 28192789
- [Background] Uberall MA, Muller-Schwefe GHH, Horlemann J. Efficacy and tolerability of the antispasmodic, pridinol, in patients with muscle-pain - results of primepain, a retrospective analysis of open-label real-world data provided by the German pain E-registry. Curr Med Res Opin. 2022 Jul;38(7):1203-1217. doi: 10.1080/03007995.2022.2077579. Epub 2022 Jun 1. PMID 35575167
- [Background] Oliveira CB, Maher CG, Pinto RZ, Traeger AC, Lin CC, Chenot JF, van Tulder M, Koes BW. Clinical practice guidelines for the management of non-specific low back pain in primary care: an updated overview. Eur Spine J. 2018 Nov;27(11):2791-2803. doi: 10.1007/s00586-018-5673-2. Epub 2018 Jul 3. PMID 29971708